CLINICAL TRIAL: NCT06927830
Title: Incidence and Risk Factors of Postoperative Nausea and Vomiting (PONV) During Elective C-Section Under Spinal Anesthesia With Multimodal Antiemetic Prophylaxis
Brief Title: Frequency of Occurrence and Risk Factors of Postoperative Nausea and Vomiting During Elective C-section Under Spinal Anesthesia With Preventive Medication
Status: Recruiting | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/534; B7072024000148 (Registry Identifier: NUB)
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Nausea and Vomiting, Postoperative; Cesarean Delivery; Spinal Anesthesia; Antiemetic Therapy
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to learn about the incidence and risk factors of nausea and vomiting during planned caesarean section under spinal anesthesia.

The main question it aims to answer is : What are the incidence and risks factors of postoperative nausea and vomiting (NV) during planned caesarean section under spinal anesthesia with administration of intrathecal morphine and multimodal antiemetic prophylaxis ?

Patients who will be managed according to the standard protocol in use in the department will have to answer specific questions about NV in the post-interventional recovery room and on 2 further visits in the first 24 hours post-caesarean section.

ELIGIBILITY:
Inclusion Criteria:

Any patient requiring elective caesarean section under spinal anesthesia, at a gestational age >37 weeks of amenorrhea in the context of a single-fetal pregnancy.

Exclusion Criteria:

Failure to understand the French language; Contraindication to locoregional anesthesia; Nausea and/or vomiting in the 24 hours preceding the procedure; Type 1 or type 2 insulin-requiring non-gestational diabetes; Allergy or contraindication to one of the products used in the usual management protocol; Severe preeclampsia; Height <150 cm

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients admitted for delivery at the CHU de Liège - Notre Dame des Bruyères site and the CHR de la Citadelle site.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of nausea and vomiting | From cesarean section to the 24th postoperative hour
  The primary endpoint will be the incidence of PONV, including the incidence of nausea requiring rescue medication; the incidence of nausea delaying resumption of oral intake (drinks, food or analgesics); and the incidence of vomiting.

SECONDARY OUTCOMES:
Risk factors of PONV | From enrollment to the 24th postoperative hour
  Risk factors will be evaluated among maternal, obstetrical, neonatal, procedural and anesthetic data.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - CHU de Liège - site de Notre-Dame des Bruyères, Chenée
  - Hôpital de la Citadelle - site Citadelle, Liège

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tan HS, Cooter M, George RB, Habib AS. A risk score for postoperative nausea and/or vomiting in women undergoing cesarean delivery with intrathecal morphine. Int J Obstet Anesth. 2020 Nov;44:126-130. doi: 10.1016/j.ijoa.2020.08.008. Epub 2020 Aug 20. PMID 32950029
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Balki M, Carvalho JC. Intraoperative nausea and vomiting during cesarean section under regional anesthesia. Int J Obstet Anesth. 2005 Jul;14(3):230-41. doi: 10.1016/j.ijoa.2004.12.004. PMID 15935649
- [Background] Sentilhes L, Schmitz T, Madar H, Bouchghoul H, Fuchs F, Garabedian C, Korb D, Nouette-Gaulain K, Pecheux O, Sananes N, Sibiude J, Senat MV, Goffinet F. [The cesarean procedure: Guidelines for clinical practice from the French College of Obstetricians and Gynecologists]. Gynecol Obstet Fertil Senol. 2023 Jan;51(1):7-34. doi: 10.1016/j.gofs.2022.10.002. Epub 2022 Oct 11. French. PMID 36228999
- [Background] Bollag L, Lim G, Sultan P, Habib AS, Landau R, Zakowski M, Tiouririne M, Bhambhani S, Carvalho B. Society for Obstetric Anesthesia and Perinatology: Consensus Statement and Recommendations for Enhanced Recovery After Cesarean. Anesth Analg. 2021 May 1;132(5):1362-1377. doi: 10.1213/ANE.0000000000005257. PMID 33177330
- [Background] Wong JY, Carvalho B, Riley ET. Intrathecal morphine 100 and 200 mug for post-cesarean delivery analgesia: a trade-off between analgesic efficacy and side effects. Int J Obstet Anesth. 2013 Jan;22(1):36-41. doi: 10.1016/j.ijoa.2012.09.006. Epub 2012 Nov 15. PMID 23159009
- [Background] Roofthooft E, Joshi GP, Rawal N, Van de Velde M; PROSPECT Working Group* of the European Society of Regional Anaesthesia and Pain Therapy and supported by the Obstetric Anaesthetists' Association. PROSPECT guideline for elective caesarean section: updated systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2021 May;76(5):665-680. doi: 10.1111/anae.15339. Epub 2020 Dec 28. PMID 33370462
- [Background] Caughey AB, Wood SL, Macones GA, Wrench IJ, Huang J, Norman M, Pettersson K, Fawcett WJ, Shalabi MM, Metcalfe A, Gramlich L, Nelson G, Wilson RD. Guidelines for intraoperative care in cesarean delivery: Enhanced Recovery After Surgery Society Recommendations (Part 2). Am J Obstet Gynecol. 2018 Dec;219(6):533-544. doi: 10.1016/j.ajog.2018.08.006. Epub 2018 Aug 15. PMID 30118692
- [Background] Van De Velde M, Vercauteren M, Stockman W, Roelants F, Coppens M, Bauters M, Ickx B, Dewandre PY, Soetens F, Cant P, Van Keer L, Gautier P. Recommendations and guidelines for obstetric anesthesia in Belgium. Acta Anaesthesiol Belg. 2013;64(3):97-104. No abstract available. PMID 24279198